CLINICAL TRIAL: NCT06089603
Title: CPAP Effect on the Polycythemia in Patients With Obstructive Sleep Apnea
Acronym: PoliAOS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Aldara García-Sánchez, M.D, pHD, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HURyC 207/23
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea, Obstructive; Polycythemia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Polycythemia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP treatment (Experimental): Diet and conventional pharmacological treatment plus continuous positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure; Drug: Conventional pharmacological treatment; Other: Sleep ,diet and life style recomendations
- Control treatment (Active Comparator): Diet and conventional pharmacological treatment
  Interventions: Drug: Conventional pharmacological treatment; Other: Sleep ,diet and life style recomendations

INTERVENTIONS:
Device: Continuous positive airway pressure — Nocturnal continuous positive airway pressure by a nasal mask. CPAP pressure will be automatically titrated using a AutoSet device (ResMed)
  Other Names: CPAP
  Arms: CPAP treatment
Drug: Conventional pharmacological treatment — Usual treatment of the patient
Other: Sleep ,diet and life style recomendations — Daily recomendatios
  Other Names: Conventional recomendations

SUMMARY:
Objectives: To compare the response of polycythemia in terms of hematocrit decrease in patients treated with positive airway pressure (CPAP) versus patients not treated with CPAP.

Methodology: Randomized, parallel-group, nonblinded, controlled clinical trial.

Patients diagnosed with OSA in a respiratory polygraphy (RP) and who meet all the inclusion criteria and none of the exclusion criteria will undergo sleepiness and quality of life questionnaires, anthropometric measurements and blood tests and will be randomized to a CPAP treatment group or control group, maintaining this treatment for 12 months. A visit will be made at 12 weeks ,24 weeks and 52 weeks to check compliance with CPAP in the treatment group and to carry out questionnaires on physical activity and quality of life, anthropometric measurements, blood tests including hemoglobin and hematocrit as well as parameters related to coagulation and platelet function and changes in medication as well as adverse effects.

Efficacy variables: blood count, hemoglobin, haematocrit, erythropoietin, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean platelet volume (MPV), platelets, coagulation, erythrocyte range of distribution (ADE), glucose, creatinine, glomerular filtration rate, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), Total bilirubin, hypoxic burden, Epworth score, EuroQol- 5D questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 18 to 80 years old.
* Diagnosis of polycytemia defined as hematocrit > 49% in men and > 48% in women. ç
* Diagnosis of moderate or severe sleep apnea, defined by an apnea-hypoapnea index >15. - Patients able to read and understand informed consent and give their signed consent.

Exclusion Criteria:

* Smokers or former smokers with pack-year index (IPA>30) or chronic obstructive pulmonary disease diagnosed by spirometry (FEV1/FVC post-bronchodilator below the lower limit of normal or z score < 1.645).
* Patients with central sleep apnea or periodic breathing
* Patients with oxygen saturation <92% or pO2< 60 mmHg at rest during wakefulness. - Evidence of severe heart failure (LVEF<50) or pulmonary hypertension.
* Patients with primary polyglobulia (polycythemia vera). It will be done prior to the inclusion in the study blood levels of erythropoietin (EPO) and determination of the mutation of the JAK2 V617F gene. Patients with normal or elevated EPO levels (normal limits 2.9- 25.9 mU/ml) and no JAK2 V617F gene mutation
* Patients with any active neoplasm will be included in the study. - Patients with chronic kidney disease (Glomerular Filtration Rate (GFR) <60 mL/min/1.73 m2).
* Patients with any active neoplasia.- Patients with chronic kidney disease (Glomerular Filtration Rate (GFR) <60 mL/min/1.73 m2).
* Need for periodic bleeding according to hematology guidelines.
* Treatment with diuretics.
* Treatment with antiplatelets or anticoagulants.
* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg at the baseline visit.
* Stroke, transient ischemic attack, acute coronary syndrome or hospitalization due to worsening heart failure, in the previous 30 days .
* Professional drivers, high-risk profession or respiratory failure (according to criteria of the clinical path of diagnosis and treatment of sleep-related respiratory disorders).
* High daytime sleepiness (Epworth sleepiness scale > 16)
* Previous treatment with CPAP- Participation in another clinical trial within 30 days prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of hematocrit | 12 months
  To compare the change in hematocrit in blood patients between the patients allocated to CPAP group and the control group

SECONDARY OUTCOMES:
Change from baseline of hemoglobin | 12 months
  To compare the change in hemoglobin in blood patients between the patients allocated to CPAP group and the control group
Change from baseline in the health-related quality of life assessed by the Euroqol-5 | 12 months
  The 5-level EQ-5D version (EQ-5D-5L) essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scal fom 0 to 100 points.
Relationship between hypoxic burden and hemoglobin and hematocrit | 12 months
  HB was defined as the total area under the oxygen saturation curve from a pre-event baseline oxygen desaturation.
  For each apnea and hypopnea the termination of the event is called "time-zero". The oxygen saturation signals around time-zero are synchronized with respect to time-zero.The time-aligned oxygen saturation signals are ensemble-averaged such that the mean value at each time point is calculated, resulting in a subject-specific average oxygen saturation curve specific to apneas and hypopneas.A subject-specific search window to quantify the area under the desaturation curve for each event is defined as the interval between the pre-event and post-event maximum oxygen saturation values. This time-locked search window will be used to determine the start and end of oxygen desaturation and calculate the area under desaturation curve for each respiratory event.Total HB (%min/h) is defined as the sum of individual areas (%min) divided by total sleep time (h).
Change from baseline in sleepiness assessed by Epworth scale | 12 months
  To compare the change in the total score and the domains of the Epworth sleepiness scale between the CPAP group and the control group.
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.
  Interpretation:
  0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24:You are excessively sleepy and should consider seeking medical attention.
Relationship between night time below SaO2 90% (T90) and oxygen desaturation index (ODI) and hematocrit | 12 months
  T90 is the percent sleep time with SpO2 below 90%. T90 measures the desaturations that dip below a threshold of 90%. Oxygen desaturation index (ODI) is the average number of desaturation episodes per hour. It is used to characterize intermittent hypoxemia (IH), an OSA-related physiological consequence that is likely responsible for most of the pathophysiological systemic complications of OSA

CONTACTS AND LOCATIONS:
Overall Officials: Aldara García-Sanchez, MD, phD, Principal Investigator — Hospital Ramon y Cajal
Locations (1):
- Aldara García-Sanchez, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No